CLINICAL TRIAL: NCT04392908
Title: Communication Memory of Cancer Diagnosis Within Pediatric Triangle: a Cross-sectional Observational Study
Brief Title: Communication Memory of Cancer Diagnosis Within the Pediatric Triangle
Status: Active, not recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Collaborators: University of Florence (Other)
Responsible Party: Principal Investigator, Rosanna Martin, Principal Investigator, Meyer Children's Hospital IRCCS
Other Study IDs: Communication in oncology
Record Dates: First submitted 2020-05-05; First posted 2020-05-19 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Memory
Keywords: memory; pediatric cancer; oncology; communication; diagnosis
MeSH Terms: conditions — Neoplasms; Communication; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients: Pediatric patients from 12 to 17 with cancer diagnosis only taken by Meyer Children's Hospital prior consent. Knowledge of fluent Italian language is required
  Interventions: Other: Communication memory
- Parents: Parents of pediatric patients prior consent. Knowledge of fluent Italian language is required
  Interventions: Other: Communication memory
- Medical Staff: Medical staff including doctor, psychologist and nurse
  Interventions: Other: Communication memory

INTERVENTIONS:
Other: Communication memory — All groups will undergo audio-recorder interviews. Only adults will complete a self-report questionnaire on phenomenological aspects of autobiographical memories.

SUMMARY:
Present project aims to investigate memories related to a cancer communication diagnosis in pediatric oncology. It evaluates possible common elements and specificity between family and healthcare staff.

DETAILED DESCRIPTION:
Lots of scientific evidences have shown that autobiographical episodes' narrative has a beneficial effect on the elaboration of memories. Indeed, narrating is a way to order thoughts and moods, which are connected to particular episodes of one's life, in order to rework and relive them. Since the diagnosis, a relationship and an open and sincere dialogue between the various parts of the pediatric triangle can promote a process of adaptation to the experience of illness and an integrated biopsychosocial healing. The first aim of this study is to explore and analyze autobiographical memories of pediatric patients, parents and healthcare staff. Also, it aims to investigate possible common and discordant element between deposition.

Phases of the present study:

1. Sample recruitment and informed consent collection.
2. Diagnosis communication audio recording.
3. Communication of the autobiographical memory of the diagnosis audio recording of patients, parents, oncologist, nurse and psychologists involved, the day after the communication.
4. Questionnaire APAM administration for adult participants.
5. Audio Transcription and data coded. Data will be registered and operated by means of statistical software as SPSS (IBM) and T-Lab (Lancia, 2004).
6. Statistical processing: ANOVA and t of Student tests will be implemented in order to compare collected questionnaires. Narrative analysis will be implemented by means of textual analysis software.

ELIGIBILITY:
Inclusion criteria for pediatric patients:

* age from 12 to 17 with cancer diagnosis only taken by Meyer Children's Hospital prior consent.
* Italian speaking

Exclusion criteria for pediatric patients:

* under 12 years old and above 17;
* followed by other hospital;
* cognitive disability

Inclusion criteria for parents:

- Italian speaking and signature informed consent.

Exclusion criteria for parents:

- cognitive disability

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with cancer diagnosis; their parents and healthcare staff
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Phenomenological characteristics of autobiographical memory | One day after diagnosis
  Self report questionnaire "Assessment of the Phenomenology of Autobiographical Memory - APAM"
Emotional characteristics of autobiographical memory | One day after diagnosis
  linguistic analysis by Linguistic Inquiry Word Count - LIWC; cluster analysis by T-Lab; Content analysis; coherence and narrative structure by High Point Anaysis.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Fioretti, PhD, Study Chair — Laboratorio di Metodi e Tecniche di Analisi delle Esperienze di Malattia Dipartimento di Scienze della Formazione e Psicologia, Università degli Studi di Firenze
Locations (1):
- Meyer Children's Hospital, Florence, Firenze, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bury M. Chronic illness as biographical disruption. Sociol Health Illn. 1982 Jul;4(2):167-82. doi: 10.1111/1467-9566.ep11339939. PMID 10260456
- [Background] Fioretti, C., & Smorti, A. (2015). How emotional content of memories changes in narrative. Narrative Inquire, 25(1), 37-56.
- [Background] Fioretti C, Smorti A. Narrating positive versus negative memories of illness: does narrating influence the emotional tone of memories? Eur J Cancer Care (Engl). 2017 May;26(3). doi: 10.1111/ecc.12524. Epub 2016 Jun 8. PMID 27271542
- [Background] Giffard B, Viard A, Dayan J, Morel N, Joly F, Eustache F. Autobiographical memory, self, and stress-related psychiatric disorders: which implications in cancer patients? Neuropsychol Rev. 2013 Jun;23(2):157-68. doi: 10.1007/s11065-013-9233-6. Epub 2013 May 3. PMID 23640242
- [Background] Habermas T, Bluck S. Getting a life: the emergence of the life story in adolescence. Psychol Bull. 2000 Sep;126(5):748-69. doi: 10.1037/0033-2909.126.5.748. PMID 10989622
- [Background] Jankovic, M. & Puricelli, E. (2008). La comunicazione della diagnosi al bambino. In S. M. G. Adamo (A cura di), La cura della relazione in oncologia pediatrica. Milano: Raffaello Cortina.
- [Background] Lancia, F. (2004). Strumenti per l'analisi dei testi: introduzione all'uso di T-Lab. Milano: Franco Angeli
- [Background] Last BF, van Veldhuizen AM. Information about diagnosis and prognosis related to anxiety and depression in children with cancer aged 8-16 years. Eur J Cancer. 1996 Feb;32A(2):290-4. doi: 10.1016/0959-8049(95)00576-5. PMID 8664044
- [Background] Levi RB, Marsick R, Drotar D, Kodish ED. Diagnosis, disclosure, and informed consent: learning from parents of children with cancer. J Pediatr Hematol Oncol. 2000 Jan-Feb;22(1):3-12. doi: 10.1097/00043426-200001000-00002. PMID 10695815
- [Background] Malterud K, Siersma VD, Guassora AD. Sample Size in Qualitative Interview Studies: Guided by Information Power. Qual Health Res. 2016 Nov;26(13):1753-1760. doi: 10.1177/1049732315617444. Epub 2016 Jul 10. PMID 26613970
- [Background] McAdams, D. P. (2008). Personal narratives and the life story. In R. John, W. Robins & L. Pervin (Eds.), Handbook of personality: Theory and Research (3rd edn, pp. 241-261). New York: Guilford Press.
- [Background] Nilsson-Ihrfelt E, Fjallskog ML, Liss A, Jakobsson O, Blomqvist C, Andersson G. Autobiographical memories in patients treated for breast cancer. J Psychosom Res. 2004 Oct;57(4):363-6. doi: 10.1016/j.jpsychores.2004.01.009. PMID 15518671
- [Background] Papini, M., Tringali, D., & Lauro-Grotto, R. (2011). La nostra era una vita normale. Ancona: Sorbello Editore.
- [Background] Parker TM, Johnston DL. Parental perceptions of being told their child has cancer. Pediatr Blood Cancer. 2008 Oct;51(4):531-4. doi: 10.1002/pbc.21667. PMID 18623217
- [Background] Pennebaker, J., Fracis, M.E., & Booth, R.J. (2001). Linquistic Inquiry Word Count: LIWC 2001. Mahway: Lawrence Erlbaum Associates.
- [Background] Smorti, A. (2007). Narrazioni. Cultura, memorie, formazione del sé. Firenze: Giunti.
- [Background] Smorti, A. & Donzelli, G.P. (2015). La medicina narrativa in pediatria. Come le storie ci aiutano a capire la malattia. Firenze: SEID.
- [Background] Sobo EJ. Good communication in pediatric cancer care: a culturally-informed research agenda. J Pediatr Oncol Nurs. 2004 May-Jun;21(3):150-4. doi: 10.1177/1043454204264408. PMID 15296044
- [Background] Tates K, Meeuwesen L. Doctor-parent-child communication. A (re)view of the literature. Soc Sci Med. 2001 Mar;52(6):839-51. doi: 10.1016/s0277-9536(00)00193-3. PMID 11234859
- [Background] Vannucci, M., Marchetti, I., Manili, A., Chiorri, C. (2010). "Come" ricordiamo il passato: Un nuovo strumento sulla fenomenologia della memoria autobiografica. Congresso Nazionale AIP; Sezione di Psicologia Sperimentale, Bologna, 2-4 Settembre 2010.
- [Background] Vannucci M, Chiorri C, Marchetti I. Shaping our personal past: Assessing the phenomenology of autobiographical memory and its association with object and spatial imagery. Scand J Psychol. 2020 Oct;61(5):599-606. doi: 10.1111/sjop.12639. Epub 2020 Apr 4. PMID 32246729